CLINICAL TRIAL: NCT07202130
Title: Investigation of The Relationship Between Upper Extremity Function in String Instrument Performers and Shoulder Proprioception, Posture, Hypermobility and Performance Anxiety
Status: Not yet recruiting | Type: Observational
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Esra, Physiotherapist, Firat University
Other Study IDs: FıratÜ-FTR-2025
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Upper Extremity Function; Shoulder Proprioception
Keywords: Hypermobility, Performance Anxiety, Shoulder Proprioception, Stringed Instrument Performer, Upper Extremity Function

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stringed Instrument Performer: musician

SUMMARY:
Work-related musculoskeletal problems are seen in many professions, including musicians. Musculoskeletal problems related to playing are defined as any weakness, numbness, pain, tingling, or other symptoms that affect a musician's ability to play a musical instrument at their usual level. Given the high workload on the upper extremities, it is likely that neurological and musculoskeletal changes and/or dysfunctions are more common in musicians. Prolonged static activity and overuse of the trunk and proximal upper extremity muscles in musicians also frequently affect upper extremity function. Nerve compression syndromes affecting the median and ulnar nerves or thoracic outlet affect many musicians. Focal dystonias seen in musicians can affect the muscles that make up part or all of one hand. Studies evaluating musculoskeletal problems and upper extremity function in instrumentalists are limited in the literature. The aim of our study is to investigate the factors affecting upper extremity function in stringed instrument performers within a group of musicians, to compare them with a group that does not play any musical instrument, and to contribute the results to the literature. A total of 68 participants will be included in the study on a voluntary basis, comprising a stringed instrument performer group (n=34) and a control group not playing any musical instrument (n=34). Upper extremity function will be assessed using the Health Throw Test, the Disability of the Arm, Shoulder, and Hand (DASH) Questionnaire and hand dynamometer, musculoskeletal system with the Nordic Musculoskeletal System Questionnaire, performance anxiety with the Kenny Music Performance Anxiety Inventory, pain with the Visual Analogue Scale (VAS), hypermobility with the Beighton Scoring System for Hypermobility and the Upper Extremity Hypermobility Questionnaire, reaction time with the Nelson Hand Reaction Test, coordination using the Touching Discs Test, posture using the Apecs-AI Posture Assessment and Correction System® (Apecs) application, shoulder proprioception using a goniometer, upper extremity balance using the Y Balance Test, and shoulder girdle endurance and stabilisation using the Closed Kinetic Chain Upper Extremity Stability Test.

DETAILED DESCRIPTION:
Work-related musculoskeletal problems are seen in many professions, including musicians. Musculoskeletal problems related to playing are defined as any weakness, numbness, pain, tingling, or other symptoms that affect a musician's ability to play a musical instrument at their usual level. Given the high workload on the upper extremities, it is likely that neurological and musculoskeletal changes and/or dysfunctions are more common in musicians. Prolonged static activity and overuse of the trunk and proximal upper extremity muscles in musicians also frequently affect upper extremity function. Nerve compression syndromes affecting the median and ulnar nerves or thoracic outlet affect many musicians. Focal dystonias seen in musicians can affect the muscles that make up part or all of one hand. Studies evaluating musculoskeletal problems and upper extremity function in instrumentalists are limited in the literature. The aim of our study is to investigate the factors affecting upper extremity function in stringed instrument performers within a group of musicians, to compare them with a group that does not play any musical instrument, and to contribute the results to the literature. A total of 68 participants will be included in the study on a voluntary basis, comprising a stringed instrument performer group (n=34) and a control group not playing any musical instrument (n=34). Upper extremity function will be assessed using the Health Throw Test, the Disability of the Arm, Shoulder, and Hand (DASH) Questionnaire and hand dynamometer, musculoskeletal system with the Nordic Musculoskeletal System Questionnaire, performance anxiety with the Kenny Music Performance Anxiety Inventory, pain with the Visual Analogue Scale (VAS), hypermobility with the Beighton Scoring System for Hypermobility and the Upper Extremity Hypermobility Questionnaire, reaction time with the Nelson Hand Reaction Test, coordination using the Touching Discs Test, posture using the Apecs-AI Posture Assessment and Correction System® (Apecs) application, shoulder proprioception using a goniometer, upper extremity balance using the Y Balance Test, and shoulder girdle endurance and stabilisation using the Closed Kinetic Chain Upper Extremity Stability Test. The relationship between the assessed parameters will be evaluated using Pearson and Spearman correlations. The Student's t-test and Mann-Whitney U test will be used for comparisons between two independent groups.

ELIGIBILITY:
Inclusion Criteria:

* Be aged between 18 and 50
* Not play any musical instrument
* Be a sedentary individual (individuals without regular exercise habits)

Exclusion Criteria:

* Being pregnant
* Having undergone surgery involving the shoulder, arm, forearm or hand region within the last 6 months
* Having any psychological diagnosis or regularly taking antidepressant medication
* Having any chronic illness that could affect upper limb function

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: musician
Sampling Method: Probability Sample
Enrollment: 68 (Estimated)
Dates: Start 2025-09-25 (Estimated); Primary Completion 2025-12-25 (Estimated); Study Completion 2026-02-05 (Estimated)

PRIMARY OUTCOMES:
upper balance assessment for musicians | From registration until the end of the assessment, 8 weeks later
  balance

SECONDARY OUTCOMES:
upper balance assessment for musicians | From registration until the end of the assessment, 8 weeks later
  balance